CLINICAL TRIAL: NCT02175212
Title: Phase III Multicenter Randomized Trial of Adjuvant Androgen Deprivation in Combination With Three-dimensional Conformal Radiotherapy Doses in High and Intermediate Risk Localized Prostate Cancer.
Brief Title: Clinical Trials of Adjuvant Androgen Deprivation in Localized Prostate Cancer
Acronym: AADLPC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fundación de Investigación Biomédica - Hospital Universitario de La Princesa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DART01/05
Record Dates: First submitted 2014-06-23; First posted 2014-06-26 (Estimated); Results first posted 2016-11-04 (Estimated); Last update posted 2020-11-20 (Actual); Status verified 2020-11

CONDITIONS: Prostate Adenocarcinoma
Keywords: Patients with prostate adenocarcinoma
MeSH Terms: interventions — Neoadjuvant Therapy; Adjuvants, Pharmaceutic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Long term androgen deprivation (Experimental): * Gosereline 3.6 mg 1 month plus 10.8 mg subcutaneously 3 months (total 4 months)
  * Bicalutamide 50 mg tablet every day for 2 months
  * High dose conformal radiotherapy
  * Gosereline 10.8 mg by subcutaneous injection every 3 moths for 2 years at the end of the radiotherapy
  Interventions: Drug: Long term androgen deprivation; Radiation: Long term androgen deprivation
- Short term androgen deprivation (Active Comparator): * Gosereline 3.6 mg 1 month plus 10.8 mg subcutaneously 3 months (total 4 months)
  * Bicalutamide 50 mg tablet every day for 2 months
  * High dose conformal radiotherapy
  Interventions: Drug: Short term androgen deprivation; Radiation: Short term androgen deprivation

INTERVENTIONS:
Drug: Short term androgen deprivation — * Gosereline 3.6 mg 1 month plus 10.8 mg subcutaneously 3 months (total 4 months)
  * Bicalutamide 50 mg tablet every day for 2 months
  Other Names: Neoadjuvant and concomitant
  Arms: Short term androgen deprivation
Drug: Long term androgen deprivation — * Gosereline 3.6 mg 1 month plus 10.8 mg subcutaneously 3 months (total 4 months)
  * Bicalutamide 50 mg tablet every day for 2 months
  * Gosereline 10.8 mg by subcutaneous injection every 3 moths for 2 years at the end of the radiotherapy
  Other Names: Neoadjuvant, concomitant and adjuvant
  Arms: Long term androgen deprivation
Radiation: Short term androgen deprivation — Minimum dose of 76 Gy (range 76-82 Gy)
  Arms: Short term androgen deprivation
Radiation: Long term androgen deprivation — Minimum dose of 76 Gy (range 76-82 Gy)
  Arms: Long term androgen deprivation

SUMMARY:
The present study is a phase III randomized and multicentric trial evaluating the potential additional impact effect of two years adjuvant androgen deprivation when combined with neoadjuvant (4 months) and high-dose (76 Gy) conformal radiotherapy in moderate high-risk prostate cancer patients. Stratification will be performed by prognostic factors and by participating institution.

ELIGIBILITY:
Inclusion Criteria:

* Histological proven adenocarcinoma of the prostate
* Stage: cT1c-3b N0M0 according to American Joint Committee on Cancer (AJCC) Tumor Node Metastasis (TNM)
* Prostatic Specific Antigen (PSA)<100 ng/ml
* Intermediate (T1-T2 with Gleason Score [GS] 7 and/or PSA 10-20)
* High risk (T3 and/or GS 8-10 and/or PSA > 20)
* Karnofsky Index (KI) performance status ≥70%
* Written informed consent

Exclusion Criteria:

* T4 N1 M1,
* Previous surgical treatment (prostatectomy or cryosurgery)
* Neoadjuvant hormonal treatment > 3 months.
* History of pelvic radiotherapy (RT)
* Contraindications for radiotherapy
* Concomitant use of chemotherapy
* Serious psychiatric or medical condition
* Current synchronic malignancies

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 362 (Actual)
Dates: Start 2005-11; Primary Completion 2014-06 (Actual); Study Completion 2020-09-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Almudena Zapatero, MD PhD, IP, Principal Investigator — Grupo de Investigación Clínica en Oncología Radioterapia
Locations (1):
- Hospital Universitario de la Princesa, Madrid, Spain

REFERENCES:
- [Background] Pollack A, Zagars GK, Starkschall G, Antolak JA, Lee JJ, Huang E, von Eschenbach AC, Kuban DA, Rosen I. Prostate cancer radiation dose response: results of the M. D. Anderson phase III randomized trial. Int J Radiat Oncol Biol Phys. 2002 Aug 1;53(5):1097-105. doi: 10.1016/s0360-3016(02)02829-8. PMID 12128107
- [Background] Zelefsky MJ, Leibel SA, Gaudin PB, Kutcher GJ, Fleshner NE, Venkatramen ES, Reuter VE, Fair WR, Ling CC, Fuks Z. Dose escalation with three-dimensional conformal radiation therapy affects the outcome in prostate cancer. Int J Radiat Oncol Biol Phys. 1998 Jun 1;41(3):491-500. doi: 10.1016/s0360-3016(98)00091-1. PMID 9635694
- [Background] Zelefsky MJ, Fuks Z, Hunt M, Lee HJ, Lombardi D, Ling CC, Reuter VE, Venkatraman ES, Leibel SA. High dose radiation delivered by intensity modulated conformal radiotherapy improves the outcome of localized prostate cancer. J Urol. 2001 Sep;166(3):876-81. PMID 11490237
- [Background] Vicini FA, Abner A, Baglan KL, Kestin LL, Martinez AA. Defining a dose-response relationship with radiotherapy for prostate cancer: is more really better? Int J Radiat Oncol Biol Phys. 2001 Dec 1;51(5):1200-8. doi: 10.1016/s0360-3016(01)01799-0. PMID 11728678
- [Background] Hanks GE, Hanlon AL, Epstein B, Horwitz EM. Dose response in prostate cancer with 8-12 years' follow-up. Int J Radiat Oncol Biol Phys. 2002 Oct 1;54(2):427-35. doi: 10.1016/s0360-3016(02)02954-1. PMID 12243818
- [Background] Leibel SA, Fuks Z, Zelefsky MJ, Hunt M, Burman CM, Mageras GS, Chui CS, Jackson A, Amols HI, Ling CC. Technological advances in external-beam radiation therapy for the treatment of localized prostate cancer. Semin Oncol. 2003 Oct;30(5):596-615. doi: 10.1016/s0093-7754(03)00354-3. PMID 14571409
- [Background] Joon DL, Hasegawa M, Sikes C, Khoo VS, Terry NH, Zagars GK, Meistrich ML, Pollack A. Supraadditive apoptotic response of R3327-G rat prostate tumors to androgen ablation and radiation. Int J Radiat Oncol Biol Phys. 1997 Jul 15;38(5):1071-7. doi: 10.1016/s0360-3016(97)00303-9. PMID 9276374
- [Background] Zietman AL, Prince EA, Nakfoor BM, Shipley WU. Neoadjuvant androgen suppression with radiation in the management of locally advanced adenocarcinoma of the prostate: experimental and clinical results. Urology. 1997 Mar;49(3A Suppl):74-83. doi: 10.1016/s0090-4295(97)00173-8. PMID 9123741
- [Background] Bolla M, Collette L, Blank L, Warde P, Dubois JB, Mirimanoff RO, Storme G, Bernier J, Kuten A, Sternberg C, Mattelaer J, Lopez Torecilla J, Pfeffer JR, Lino Cutajar C, Zurlo A, Pierart M. Long-term results with immediate androgen suppression and external irradiation in patients with locally advanced prostate cancer (an EORTC study): a phase III randomised trial. Lancet. 2002 Jul 13;360(9327):103-6. doi: 10.1016/s0140-6736(02)09408-4. PMID 12126818
- [Background] Pilepich MV, Winter K, John MJ, Mesic JB, Sause W, Rubin P, Lawton C, Machtay M, Grignon D. Phase III radiation therapy oncology group (RTOG) trial 86-10 of androgen deprivation adjuvant to definitive radiotherapy in locally advanced carcinoma of the prostate. Int J Radiat Oncol Biol Phys. 2001 Aug 1;50(5):1243-52. doi: 10.1016/s0360-3016(01)01579-6. PMID 11483335
- [Background] Lawton CA, Winter K, Murray K, Machtay M, Mesic JB, Hanks GE, Coughlin CT, Pilepich MV. Updated results of the phase III Radiation Therapy Oncology Group (RTOG) trial 85-31 evaluating the potential benefit of androgen suppression following standard radiation therapy for unfavorable prognosis carcinoma of the prostate. Int J Radiat Oncol Biol Phys. 2001 Mar 15;49(4):937-46. doi: 10.1016/s0360-3016(00)01516-9. PMID 11240234
- [Background] Granfors T, Modig H, Damber JE, Tomic R. Combined orchiectomy and external radiotherapy versus radiotherapy alone for nonmetastatic prostate cancer with or without pelvic lymph node involvement: a prospective randomized study. J Urol. 1998 Jun;159(6):2030-4. doi: 10.1016/S0022-5347(01)63235-X. PMID 9598512
- [Background] Zagars GK, Johnson DE, von Eschenbach AC, Hussey DH. Adjuvant estrogen following radiation therapy for stage C adenocarcinoma of the prostate: long-term results of a prospective randomized study. Int J Radiat Oncol Biol Phys. 1988 Jun;14(6):1085-91. doi: 10.1016/0360-3016(88)90383-5. PMID 3133327
- [Background] Pilepich MV, Winter K, Lawton CA, Krisch RE, Wolkov HB, Movsas B, Hug EB, Asbell SO, Grignon D. Androgen suppression adjuvant to definitive radiotherapy in prostate carcinoma--long-term results of phase III RTOG 85-31. Int J Radiat Oncol Biol Phys. 2005 Apr 1;61(5):1285-90. doi: 10.1016/j.ijrobp.2004.08.047. PMID 15817329
- [Background] Jani AB, Basu A, Abdalla I, Connell PP, Krauz L, Vijayakumar S. Impact of hormone therapy when combined with external beam radiotherapy for early-stage, intermediate-, or high-risk prostate cancer. Am J Clin Oncol. 2003 Aug;26(4):382-5. doi: 10.1097/01.COC.0000026483.80660.94. PMID 12902891
- [Background] Nguyen KH, Horwitz EM, Hanlon AL, Uzzo RG, Pollack A. Does short-term androgen deprivation substitute for radiation dose in the treatment of high-risk prostate cancer? Int J Radiat Oncol Biol Phys. 2003 Oct 1;57(2):377-83. doi: 10.1016/s0360-3016(03)00573-x. PMID 12957248
- [Result] Zapatero A, Valcarcel F, Calvo FA, Algas R, Bejar A, Maldonado J, Villa S. Risk-adapted androgen deprivation and escalated three-dimensional conformal radiotherapy for prostate cancer: Does radiation dose influence outcome of patients treated with adjuvant androgen deprivation? A GICOR study. J Clin Oncol. 2005 Sep 20;23(27):6561-8. doi: 10.1200/JCO.2005.09.662. PMID 16170164
- [Derived] Zapatero A, Guerrero A, Maldonado X, Alvarez A, San-Segundo CG, Rodriguez MAC, Sole JM, Olive AP, Casas F, Boladeras A, de Vidales CM, de la Torre MLV, Vara S, Sanz JL, Calvo FA. High-dose radiotherapy and risk-adapted androgen deprivation in localised prostate cancer (DART 01/05): 10-year results of a phase 3 randomised, controlled trial. Lancet Oncol. 2022 May;23(5):671-681. doi: 10.1016/S1470-2045(22)00190-5. Epub 2022 Apr 12. PMID 35427469
- [Derived] Zapatero A, Guerrero A, Maldonado X, Alvarez A, Gonzalez-San Segundo C, Cabeza Rodriguez MA, Macias V, Pedro Olive A, Casas F, Boladeras A, Martin de Vidales C, Vazquez de la Torre ML, Calvo FA. Late Radiation and Cardiovascular Adverse Effects After Androgen Deprivation and High-Dose Radiation Therapy in Prostate Cancer: Results From the DART 01/05 Randomized Phase 3 Trial. Int J Radiat Oncol Biol Phys. 2016 Oct 1;96(2):341-348. doi: 10.1016/j.ijrobp.2016.06.2445. Epub 2016 Jun 22. PMID 27598804
- [Derived] Zapatero A, Guerrero A, Maldonado X, Alvarez A, Gonzalez San Segundo C, Cabeza Rodriguez MA, Macias V, Pedro Olive A, Casas F, Boladeras A, de Vidales CM, Vazquez de la Torre ML, Villa S, Perez de la Haza A, Calvo FA. High-dose radiotherapy with short-term or long-term androgen deprivation in localised prostate cancer (DART01/05 GICOR): a randomised, controlled, phase 3 trial. Lancet Oncol. 2015 Mar;16(3):320-7. doi: 10.1016/S1470-2045(15)70045-8. Epub 2015 Feb 19. PMID 25702876

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between Nov 7, 2005, and Dec 20, 2010, 362 were registered. Of these, seven did not meet the inclusion criteria. The final trial population thus consisted of 355 men, of whom 178 were randomly assigned to the short-term androgen deprivation group and 177 to the long-term androgen deprivation group.
Groups:
- Long Term Androgen Deprivation: * Gosereline 3.6 mg 1 month plus 10.8 mg subcutaneously 3 months (total 4 months)
  * Bicalutamide 50 mg tablet every day for 2 months
  * High dose conformal radiotherapy
  * Gosereline 10.8 mg by subcutaneous injection every 3 moths for 2 years at the end of the radiotherapy
  Long term androgen deprivation: - Gosereline 3.6 mg 1 month plus 10.8 mg subcutaneously 3 months (total 4 months)
  * Bicalutamide 50 mg tablet every day for 2 months
  * Gosereline 10.8 mg by subcutaneous injection every 3 moths for 2 years at the end of the radiotherapy
  Long term androgen deprivation: Minimum dose of 76 Gy (range 76-82 Gy)
- Short Term Androgen Deprivation: * Gosereline 3.6 mg 1 month plus 10.8 mg subcutaneously 3 months (total 4 months)
  * Bicalutamide 50 mg tablet every day for 2 months
  * High dose conformal radiotherapy
  Short term androgen deprivation: - Gosereline 3.6 mg 1 month plus 10.8 mg subcutaneously 3 months (total 4 months)
  - Bicalutamide 50 mg tablet every day for 2 months
  Short term androgen deprivation: Minimum dose of 76 Gy (range 76-82 Gy)
Period: Overall Study
Arm/Group | Long Term Androgen Deprivation | Short Term Androgen Deprivation
Started | 177 | 178
Completed | 14 | 31
Not Completed | 163 | 147

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Long Term Androgen Deprivation | Short Term Androgen Deprivation | Total
Number analyzed (Participants) | 177 | 178 | 355
Age, Continuous [Median (Full Range); unit: Years] | 71 [56 to 82] | 72 [54 to 85] | 71 [54 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 177 | 178 | 355
Risk subgroup (intermediate vs. high) [Number; unit: participants]
  Intermediate | 85 | 81 | 166
  High | 92 | 97 | 189
T stage (categorical) [Number; unit: participants] — Patients were staged according to the AJCC Cancer Staging criteria, 6th edition. Intermediate-risk and high-risk factors were defined following the 2005 guidelines of the National Comprehensive Cancer Network.
  participants
    T1: tumor neither palpable not visible by imaging | 38 | 42 | 80
    T2: Tumor confinent whitin prostate | 100 | 103 | 203
    T3: Tumor extends through the prostate capsule | 39 | 33 | 72
PSA (continous) [Median (Full Range); unit: nanogrames per milliliter (ng/mL)] | 11.1 [3.1 to 72.0] | 11.0 [3.4 to 66.0] | 11 [3.1 to 72.0]
PSA (categorical) [Number; unit: participants]
  <10 ng/mL | 80 | 74 | 154
  10-20 ng/mL | 61 | 64 | 125
  >20 ng/mL | 36 | 40 | 76
Gleason score (categorical) [Number; unit: participants] — Gleason classification for prostate cancer were used considering Gleason 6 as less aggressive and Gleason 10 most aggressive
  participants
    <=6 | 21 | 30 | 51
    7 | 110 | 103 | 213
    8-10 | 46 | 45 | 91
Positive biopsy samples (continous) [Median (Full Range); unit: number of cylindres] | 4 [1 to 13] | 4 [1 to 16] | 4 [1 to 16]
Prostate radiotherapy dose (continous) [Median (Full Range); unit: Grays (Gy)] | 78.0 [30.6 to 88.4] | 78.0 [64.0 to 82.2] | 78.0 [30.6 to 88.4]
Prostate radiotherapy dose (categorical) [Number; unit: participants] — 173 evaluable patients in short term group and 171 in the long term group
  participants
    <78 Gy | 43 | 51 | 94
    >= 78 Gy | 128 | 122 | 250
Pelvic radiotherapy (categorical) [Number; unit: participants] — 173 evaluable patients in short term group and 171 in the long term group
  participants
    Yes | 20 | 28 | 48
    No | 148 | 145 | 293
    Missing | 3 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Biochemical Disease Free Survival: Estimated Percentage of Participants With Biochemical Disease-free Survival at 5 Years
Description: Biochemical relapse was defined as the time from inclusion in the study (randomization) until the patient meets criteria for Biochemical failure (Phoenix criteria: PSA nadir plus 2 ng/ml).
Time Frame: 5 years
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Long Term Androgen Deprivation | Short Term Androgen Deprivation
Number analyzed (Participants) | 177 | 178
percentage of patients | 90 [87 to 92] | 81 [78 to 81]
Statistical Analysis 1: Comparison: Long Term Androgen Deprivation vs Short Term Androgen Deprivation; Test type: Superiority or Other; p = 0.01, Regression, Cox; Hazard Ratio (HR) = 1.88, 95% CI 2-sided [1.12 to 3.15]

2. Secondary Outcome: Metastasis Free Survival: Estimated Percentage of Participants With Metastasis-free Survival at 5 Years
Description: Metastasis free survival: defined as the time from inclusion in the study (randomization) until the appearance of distant metastases: a positive result in any of the tests performed (scintigraphy, chest radiography, thorax, abdominal and pelvic CT and MRI).
Time Frame: 5 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Long Term Androgen Deprivation | Short Term Androgen Deprivation
Number analyzed (Participants) | 177 | 178
percentage of participants | 94 [92 to 96] | 83 [80 to 86]
Statistical Analysis 1: Comparison: Long Term Androgen Deprivation vs Short Term Androgen Deprivation; Test type: Superiority or Other; p = 0.01, Regression, Cox; Hazard Ratio (HR) = 2.31, 95% CI 2-sided [1.23 to 3.85]

3. Secondary Outcome: Overall Survival: Estimated Percentage of Participants Alive at 5 Years
Description: Overall Survival: defined as the time that elapses from the patient enters the study until the patient dies from any cause.
Time Frame: 5 years
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Long Term Androgen Deprivation | Short Term Androgen Deprivation
Number analyzed (Participants) | 177 | 178
percentage of patients | 95 [93 to 97] | 86 [83 to 89]
Statistical Analysis 1: Comparison: Long Term Androgen Deprivation vs Short Term Androgen Deprivation; Test type: Superiority or Other; p = 0.009, Regression, Cox; Hazard Ratio (HR) = 2.48, 95% CI 2-sided [1.31 to 4.68]

4. Secondary Outcome: Cause-specific Survival
Description: Cause-specific survival included all deaths from prostate cancer or treatment complications, and deaths from unknown causes in patients with either active cancer or a previously documented relapse
Time Frame: 5 years
Measure: Number; unit: participants
Arm/Group | Long Term Androgen Deprivation | Short Term Androgen Deprivation
Number analyzed (Participants) | 177 | 178
participants | 177 | 173

5. Secondary Outcome: Late Toxicity
Description: Defined as the maximal rectal, urinary and cardiovascular (CV) toxicity per patient more than 90 days after completion of RT.
  Scoring scales used were the radiation morbidity scoring criteria of the European Organization for Research and Treatment of Cancer-Radiation Therapy Oncology Group (EORTC/RTOG) and the Common Terminology Criteria for Adverse Events (CTCAEs) v 3.0 for the remained toxicity.
  CV events were defined according to the World Health Organization criteria
Time Frame: 5 years
Measure: Number; unit: percentage of patients
Arm/Group | Long Term Androgen Deprivation | Short Term Androgen Deprivation
Number analyzed (Participants) | 177 | 178
percentage of patients
  Grade 2 of more rectal toxicity | 11.1 | 7.6
  Grade 2 of more urinary toxicity | 8.2 | 7.3
  Cardiovascular | 17.6 | 7.2

ADVERSE EVENTS:
Time Frame: 63 months (IQR 50-82)
Description: Maximum toxicity per patient
Arm/Group | Long Term Androgen Deprivation | Short Term Androgen Deprivation
Serious Adverse Events (participants affected / at risk) | 36/177 | 29/178
Other Adverse Events (participants affected / at risk) | 62/177 | 40/178
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Long Term Androgen Deprivation (N=177) | Short Term Androgen Deprivation (N=178)
Miocardial Infarction/Ischemic disease (Cardiac disorders) | 11 (11) | 4 (4)
Tromboembolic disease (Vascular disorders) | 4 (4) | 4 (4)
Cerebrovascular accident (CVA) (Vascular disorders) | 5 (5) | 3 (3)
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Second malignancies (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 12 (12) | 14 (15)
Sepsis (Infections and infestations) | 2 (2) | 4 (4)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Long Term Androgen Deprivation (N=177) | Short Term Androgen Deprivation (N=178)
Rectal bleeding (Gastrointestinal disorders) | 12 (12) | 14 (14) — Grade 2 or more according EORTC/RTOG and CTCAE v 3.0
Urinary toxicity (Renal and urinary disorders) | 9 (9) | 10 (10) — Grade 2 or more according EORTC/RTOG and CTCAE v 3.0
Asthenia (General disorders) | 13 (13) | 3 (3)
Hot flashes (Metabolism and nutrition disorders) | 28 (28) | 13 (13) — Grade 2 or more according EORTC/RTOG and CTCAE v 3.0

LIMITATIONS AND CAVEATS:
* Relatively short follow-up and low number of events.
* The lack of patient-reported outcomes.
* Our decision to include vascular events other than strictly cardiac events (e.g. the presence of CVA or thromboembolic disease).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No